CLINICAL TRIAL: NCT05103384
Title: Utilizing Neural Signatures and Virtual Reality to Advance DBS Programming
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Principal Investigator, Jay Alberts, Principal Investigator; Staff, Biomedical Engineering, The Cleveland Clinic
Other Study IDs: 21-957
Record Dates: First submitted 2021-09-30; First posted 2021-11-02 (Actual); Results first posted 2025-11-04 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-08

CONDITIONS: Parkinson Disease; DBS; Deep Brain Stimulation; Freezing of Gait; Virtual Reality
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- PD Virtual Reality Cohort
  Interventions: Other: Virtual Reality Environment

INTERVENTIONS:
Other: Virtual Reality Environment — Participants complete various tasks in a virtual home and grocery store environment.

SUMMARY:
The project uses virtual reality technology to recreate situations that cause freezing of gait in individuals with Parkinson's disease. Individuals who underwent deep brain stimulator (DBS) surgery for Parkinson's disease will walk through a virtual reality environment while brain signals are recorded from the DBS device. The goal is to better understand what occurs in the brain during freezing of gait.

DETAILED DESCRIPTION:
Falls related to problems with posture and walking as well as freezing of gait (FOG) occur in nearly 80% of people with Parkinson's disease (PD). Despite falls occurring in the daily lives of people with PD, it is difficult to produce FOG episodes in a doctor's office or other clinical setting. We will therefore use virtual reality to create an environment that can consistently produce FOG episodes in people with PD. By purposely producing FOG while people are wearing equipment that monitors brain activity, we can see where in the brain FOG is triggered. Study participants will be asked to wear a virtual reality (VR) headset and heart rate monitor and walk on a treadmill that permits users to start, stop, and turn, allowing them to naturally walk through a virtual environment. We will record the activity from the DBS system while participants perform the tasks. Participants will also complete clinical assessments of PD, a FOG questionnaire and cognitive tests that include naming objects and recalling items from a list.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of idiopathic PD
* Undergoing scheduled surgery for bilateral STN-DBS at a Cleveland Clinic facility or previously undergone STN-DBS surgery with the Medtronic Percept BrainSense DBS system
* Self-reported response of one or greater on question #3 of the Freezing of Gait Questionnaire (FOG-Q)
* Ability to walk independently for a minimum of 10 minutes
* Ability to provide informed consent

Exclusion Criteria:

* Neurological disease other than PD, such as stroke or multiple sclerosis
* Musculoskeletal impairment that affects one's ability to ambulate
* Presence of active and untreated psychiatric symptoms meeting Diagnostic and Statistical Manual of Mental Disorders-4th Edition (DSM-IV) criteria for Axis-I disorder. Depression and anxiety are very common in patients with Parkinson's disease and are often mitigated as part of routine care. Depression and anxiety will not preclude study participation
* Cognitive impairment meeting Diagnostic and Statistical Manual of Mental Disorders-4th Edition (DSM-IV) criteria for dementia on formal neuropsychological evaluation
* Current alcohol or substance abuse
* Hearing or visual impairment precluding VR use
* Lack of fluency in English which may invalidate certain tests

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson's disease undergoing bilateral STN-DBS surgery at a Cleveland Clinic Facility or who have previously undergone STN-DBS surgery with the Medtronic Percept BrainSense DBS system.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2022-07-22 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay Alberts, Ph.D., Principal Investigator — Staff
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- PD Virtual Reality Cohort: Participants with Parkinson's disease complete cognitive and motor tasks while wearing a virtual reality headset and walking on an omnidirectional treadmill. The virtual reality headset immerses the participant in a virtual home environment designed to elicit freezing of gait episodes. While completing tasks in the virtual home environment, researchers monitor for freezing of gait episodes to investigate neural signatures associated with freezing. Each participant completed the virtual reality modules under two conditions: OFF DBS/OFF PD Meds and OFF DBS/ON PD Meds.
Period: Overall Study
Arm/Group | PD Virtual Reality Cohort
Started | 15
Completed | 11
Not Completed | 4
Not completed — Too severely affected Off Meds/Off DBS to complete entire protocol | 4

BASELINE CHARACTERISTICS:
Arm/Group | PD Virtual Reality Cohort
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.8 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11
Parkinson's Disease Duration [Mean (Standard Deviation); unit: years] | 10.1 (5.1)
Years since DBS Placement [Mean (Standard Deviation); unit: years] | 2.5 (3.7)
MDS-UPDRS III, OFF MEDS/OFF DBS [Mean (Standard Deviation); unit: score on a scale] — Global score of motor function in Parkinson's disease using the Movement Disorders Society-Unified Parkinson's Disease Rating Scale subscale III (MDS-UPDRS III). Eighteen items scored on a 0-4 scale resulting in a combined score ranging from 0-72. A higher score (larger number) indicates more motor symptoms.
  score on a scale | 59.2 (19.7)

OUTCOME MEASURES:

1. Primary Outcome: Freezing of Gait
Description: Number of freezing of gait episodes
Time Frame: Baseline
Population: Participants were assessed in the Off DBS/Off Meds condition and Off DBS/On Meds condition for outcome measures. No other conditions were assessed.
Measure: Mean (Standard Deviation); unit: freezing of gait episodes
Groups:
- OFF DBS/OFF PD Meds: Session completed with DBS stimulation turned off and participant off their PD meds for 12 hours prior. All analyzed participants completed a session OFF DBS/OFF PD Meds and OFF DBS/ON Meds.
- OFF DBS/ON PD Meds: Session completed with DBS stimulation turned off and participant on their PD meds. All analyzed participants completed a session OFF DBS/OFF PD Meds and OFF DBS/ON Meds.
Arm/Group | OFF DBS/OFF PD Meds | OFF DBS/ON PD Meds
Number analyzed (Participants) | 11 | 11
freezing of gait episodes | 2.6 (2.6) | 1.5 (2.1)

2. Secondary Outcome: Gait Velocity
Description: Meters/second
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | OFF DBS/OFF PD Meds | OFF DBS/ON PD Meds
Number analyzed (Participants) | 11 | 11
m/s | 0.27 (0.06) | 0.29 (0.07)

3. Secondary Outcome: Turn Velocity
Description: Degrees/second
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: degrees/s
Arm/Group | OFF DBS/OFF PD Meds | OFF DBS/ON PD Meds
Number analyzed (Participants) | 11 | 11
degrees/s | 21.7 (6.0) | 22.1 (5.9)

ADVERSE EVENTS:
Time Frame: Through study completion, which was an average of 1 week.
Groups:
- Off DBS/Off Meds: Session completed with DBS stimulation turned off and participant OFF their PD meds for 12 hours prior.
- Off DBS/On Meds: Session completed with DBS stimulation turned off and participant ON their PD meds.
Arm/Group | Off DBS/Off Meds | Off DBS/On Meds
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 1/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Off DBS/Off Meds (N=15) | Off DBS/On Meds (N=15)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-27): https://cdn.clinicaltrials.gov/large-docs/84/NCT05103384/Prot_SAP_000.pdf